CLINICAL TRIAL: NCT02005614
Title: A Pilot/Phase II Study of Gamma Knife Radiosurgery for Brain Metastases Using 3Tesla MRI and Rational Dose Selection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit patients.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1306012291
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Melanoma; Renal Cell Carcinoma; Sarcoma; Breast Cancer; Lung Cancer; Colorectal Cancer; Gastrointestinal Cancers; Brain Metastases
Keywords: Rational dose selection; gamma knife radiosurgery
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Sarcoma; Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Gastrointestinal Neoplasms; Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gamma Knife Radiosurgery (Experimental): "Rational dose selection" is a concept wherein doses used for stereotactic radiosurgery is selected based on tumor volume, prior irradiation with whole brain radiotherapy, and the relative radioresistance of the tumor (radioresistant = melanoma, renal cell carcinoma, sarcoma; radiosensitive = breast cancer, lung cancer, colorectal cancer, gastrointestinal cancers).
  Dose may be altered for lesions in the brainstem, adjacent to the optic nerve, optic chiasm, or motor cortex, or other clinical scenarios as defined by the treating physician. Reason for dose alteration will be recorded at the time of treatment.
  For patients with 10+ brain metastases with multimorbidity or difficulty in tolerating a supine position, doses may be modified by the treating physicians for patient comfort.
  Interventions: Procedure: Gamma Knife Radiosurgery

INTERVENTIONS:
Procedure: Gamma Knife Radiosurgery — Treatment will be administered on an outpatient basis. No other treatment, investigational or commercial agents or therapies other than those described below may be administered with the intent to treat the patient's brain metastases.
  Gamma knife radiosurgery is a one day out-patient procedure. Time from initiation of treatment (premedication and placement of a stereotactic frame) until end of treatment (completion of radiation delivery and removal of stereotactic frame) ranges from 3 to 16 hours.

SUMMARY:
The purpose of this study is to collect prospective data for use as a comparator for future subsequent studies attempting to increase the efficacy or reduce the toxicity of gamma knife radiosurgery.

DETAILED DESCRIPTION:
The aims of this study are to pilot a study to measure local control after "rational dose" selected gamma knife radiosurgery for brain metastases and to measure treatment related toxicity for rational dose selected gamma knife radiosurgery for brain metastases. In addition, the quality of life and neurocognition of patients undergoing gamma knife radiosurgery will be measured using the validated European Organisation for Research and Treatment of Cancer QLQ-C30 and QLQ-BN20 survey instruments. "Rational dose selection" is a concept wherein doses used for stereotactic radiosurgery is selected based on tumor volume, prior irradiation with whole brain radiotherapy, and the relative radioresistance of the tumor (radioresistant = melanoma, renal cell carcinoma, sarcoma; radiosensitive = breast cancer, lung cancer, colorectal cancer, gastrointestinal cancers).

Eligible patients will have histologically confirmed cancer and MRI evidence of metastatic disease within the brain. Patients will be eligible for the trial if intracranial radiosurgery has been recommended for treatment of brain metastases. Patients will be excluded if they have an extremely radiosensitive tumor (leukemia, lymphoma), a radiosensitivity syndrome, a resection of a brain metastasis, or cannot tolerate the MRI or placement of a stereotactic head frame. All patients must sign informed consent.

Radiation will consist of gamma knife radiosurgery delivered using doses selected based on the concept of "rational dose selection" as summarized above.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed malignancy (not leukemia or lymphoma). There must be metastatic brain disease apparent on magnetic resonance imaging which offers a medical indication for brain radiation. - Age > 18
* Karnofsky Performance Status > 70
* MRI performed within 4 weeks of trial enrollment
* Medical oncologist or consenting physician verifies that chemotherapy options exist after treatment with intracranial therapy, and that chemotherapy is planned to initiate after completion of radiation. Or, survival as estimated by the medical oncologist or enrolling physician is > 3 months.

Exclusion Criteria:

* Extremely radiosensitive tumor (lymphoma, leukemia)
* Radiosensitivity syndrome (scleroderma, dermatomyositis, other genetic syndrome that predisposes to adverse radiotherapy complications)
* Evidence of leptomeningeal dissemination
* Resection of brain metastases, otherwise untreated with radiation for those brain lesions (presenting for postoperative consolidative radiotherapy)
* Presence of a medical device (pacemaker, stent) or allergy that precludes contrast enhanced MRI
* Patient is unable to tolerate placement of a stereotactic headframe
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-11; Primary Completion 2018-02 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Rate of Local Control Over time (RECIST Criteria) | Up to 2 years
  Response or progression of the radiated lesion will be measured by change in the largest unidimensional measurement.
  Additionally, response and progression will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee
  Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria. Local control is defined as a lack of progressive disease, as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria of a 20% increase in the longest diameter for a target lesion.
  If the lesion grows beyond 20% of the longest diameter of the pre-treatment, but subsequently regresses without further lesion-targeted radiotherapy, it will be assumed that the lesion was treatment related radiation necrosis in analysis

CONTACTS AND LOCATIONS:
Overall Officials: James B Yu, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States